CLINICAL TRIAL: NCT05566132
Title: Preventive Norepinephrine Infusion During Surgery for Upper Femoral Fracture and Post-operative Acute Renal Failure
Acronym: NORAKI
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: NORAKI
Record Dates: First submitted 2022-09-30; First posted 2022-10-04 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Femur Fracture; Acute Renal Failure
MeSH Terms: conditions — Femoral Fractures; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The fracture of the upper extremity of the femur (FESF) is one of the most common fractures in traumatology. In France, FESF affects more than 65,000 individuals per year and could involve up to 150,000 people per year by 2050, due to the increase in life expectancy of the population. The main risk factors for the occurrence of ESF are: age, gender, osteoporosis, undernutrition, gait and balance disorders. The main risk factors for death identified by the French Society of Orthopaedic Surgery and Geriatrics after surgery for ESF are: a delay between the trauma and surgery of more than 48 hours, poorly tolerated preoperative anemia or a hemoglobinemia of less than 8 g/dl, absence of antibiotic prophylaxis, postoperative acute renal failure, and discontinuation of antiaggregant treatments in the case of coronary disease. Post-operative Acute Kidney Injury (AKI) is one of the risk factors for mortality after surgery for ESF. AKI is an impairment of normal kidney function, and in general, AKI is a major issue in the management of patients undergoing surgery. In the short term, it increases the length of stay of patients, and the number of admissions to continuing care. AKI increases post-operative mortality by more than 50%. However, because of the complications associated with vascular filling, the use of vasoconstrictor drugs, such as ephedrine, phenylephrine, and especially norepinephrine, is increasingly common. Compared with other catecholamines, norepinephrine has been shown to be more effective in increasing cardiac output. Moreover, unlike bolus administration of ephedrine or phenylephrine, which favor the occurrence of blood pressure peaks and valleys, norepinephrine, administered as a continuous infusion, allows blood pressure to be maintained in a narrower range. The challenge is to implement a strategy to reduce their frequency. Intraoperative arterial hypotension is one of the risk factors on which investigators can intervene thanks to the "preventive" administration of noradrenaline in continuous infusion, started before or immediately after the induction of anesthesia. However, the "preventive" use of norepinephrine may favor the occurrence of AKI in hypovolemic patients (fracture and surgery-related bleeding, prolonged fasting) by reducing renal blood flow. Our primary objective is to compare the risk of AKI occurrence during a "preventive" norepinephrine administration strategy with a target MAP ≥65 mmHg compared with that observed in response to a vasoconstrictor-only administration strategy in response to the occurrence of arterial hypotension episodes. Secondary objectives are to evaluate the potential interactions of this preventive strategy with other risk factors for postoperative AKI.

ELIGIBILITY:
Inclusion Criteria:

* Patient 18 years of age or older
* Patient hospitalized for a fracture of the upper end of the femur
* French speaking patient

Exclusion Criteria:

* Patient with severe or end-stage chronic renal disease preoperatively
* Patient with no anesthesia report in DxCare®.
* Patient who does not have an ICU report in DxCare®.
* Patients who did not have a creatinine measurement in the emergency room or in the postoperative period
* Patients who did not receive vasoconstrictors during surgery
* Patients who tested positive for, or were diagnosed with, SARS-COV 2 infection
* Patients under guardianship or curatorship
* Patient deprived of liberty
* Patient under court protection
* Patients who object to the use of their medical data in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: - Patient 18 years of age or older, hospitalized for a fracture of the upper end of the femur.
Sampling Method: Non-Probability Sample
Enrollment: 676 (Actual)
Dates: Start 2022-08-09 (Actual); Primary Completion 2022-09-09 (Actual); Study Completion 2023-09-11 (Actual)

PRIMARY OUTCOMES:
Risk of acute renal failure with a "preventive" norepinephrine administration strategy | Day 2
  This outcome corresponds to the incidence of acute renal failure defined as an increase in postoperative creatinine value to 1.5 times baseline or an increase of 26.5 mmol/L in blood creatinine from baseline.

SECONDARY OUTCOMES:
Effect of the two strategies according to preoperative/operative risk factors | Day 2
  This outcome corresponds to the presence/absence of preoperative risk factors

CONTACTS AND LOCATIONS:
Overall Officials: Pascal ALFONSI, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, France

REFERENCES:
- [Background] Bhandari M, Swiontkowski M. Management of Acute Hip Fracture. N Engl J Med. 2017 Nov 23;377(21):2053-2062. doi: 10.1056/NEJMcp1611090. No abstract available. PMID 29166235
- [Background] Brauer CA, Coca-Perraillon M, Cutler DM, Rosen AB. Incidence and mortality of hip fractures in the United States. JAMA. 2009 Oct 14;302(14):1573-9. doi: 10.1001/jama.2009.1462. PMID 19826027
- [Background] Dadure C, Marie A, Seguret F, Capdevila X. One year of anaesthesia in France: A comprehensive survey based on the national medical information (PMSI) database. Part 1: In-hospital patients. Anaesth Crit Care Pain Med. 2015 Aug;34(4):191-7. doi: 10.1016/j.accpm.2014.12.003. Epub 2015 Jun 30. PMID 26141685
- [Background] Sykes L, Kalra PA, Green D. Comparison of impact on death and critical care admission of acute kidney injury between common medical and surgical diagnoses. PLoS One. 2019 Apr 11;14(4):e0215105. doi: 10.1371/journal.pone.0215105. eCollection 2019. PMID 30973921
- [Background] Ahuja S, Mascha EJ, Yang D, Maheshwari K, Cohen B, Khanna AK, Ruetzler K, Turan A, Sessler DI. Associations of Intraoperative Radial Arterial Systolic, Diastolic, Mean, and Pulse Pressures with Myocardial and Acute Kidney Injury after Noncardiac Surgery: A Retrospective Cohort Analysis. Anesthesiology. 2020 Feb;132(2):291-306. doi: 10.1097/ALN.0000000000003048. PMID 31939844
- [Background] Wood RJ, White SM. Anaesthesia for 1131 patients undergoing proximal femoral fracture repair: a retrospective, observational study of effects on blood pressure, fluid administration and perioperative anaemia. Anaesthesia. 2011 Nov;66(11):1017-22. doi: 10.1111/j.1365-2044.2011.06854.x. Epub 2011 Aug 18. PMID 21851345